CLINICAL TRIAL: NCT01081015
Title: Connect™ CLL: The Chronic Lymphocytic Leukemia Disease Registry
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: Connect™ CLL
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; disease registry; Connect™
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the Connect™ Chronic Lymphocytic Leukemia (CLL) Disease Registry is to explore the history and real world management of patients diagnosed with CLL, provide insight into the management of CLL, and evaluate the effectiveness of first, second and subsequent therapeutic strategies employed in both the community and academic settings.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis with CLL
* Clinical decision made to initiate first-line therapy, second-line therapy or subsequent line of therapy prior to enrollment into the ConnectTM CLL registry, but within 2 months of enrollment
* Age≥18 years
* Willing and able to provide signed informed consent
* Willing and able to complete patient assessment questionnaires either alone or with minimal assistance from caregivers and/or trained site personnel

Exclusion Criteria:

* Participation in a clinical study in which study treatment is blinded
* Patient condition is considered terminal (i.e.<6 months to live)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An adult population (>=18 years old) of both men and women who have chronic lymphocytic leukemia treated in either community or academic medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 1494 (Actual)
Dates: Start 2010-03-19 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Identify and summarize patterns in therapeutic regimens and patient outcomes | up to 8 years
  The primary objective is to 1) describe practice patterns of first line therapy regimens and subsequent therapeutic strategies in patients initiated on therapy for CLL, as well as initiated on second line and subsequent therapies, in the community and academic setting (2) Provide insight into therapeutic regimens and therapy sequence in clinical practice as they relate to clinical outcomes in patients initiated on first-line, second-line or subsequent therapies for CLL.

SECONDARY OUTCOMES:
Summarize Effectiveness of Treatment Regimens | up to 8 years
  Describe any differences in effectiveness associated with treatment regimens, including first-line regimens and subsequent therapeutic strategies in patients actively treated for CLL
Health Related Quality of Life Measures Related to Therapeutic Regimens | up to 8 years
  Describe the health-related quality of life of patients actively treated for CLL, and to explore the association of HRQoL with therapeutic regimens, sequences and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Foon, MD, Study Director — Celgene Corporation
Locations (165):
- United States (165):
  - New Hope Cancer & Research Institute, Pomona, California
  - Medical Specialists of the Palm Beaches, Atlantis, Florida
  - University Cancer Institute, Boynton Beach, Florida
  - Thomas Niederman, MD, Boynton Beach, Florida
  - Pasco Hernando Oncology Associates (Kumar), New Port Richey, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Peachtree Hematology-Oncology Consultants, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - US Oncology - Dublin Hematology & Oncology, Dublin, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - US Oncology - Cancer Care & Hematology Specialists of Chicagoland - Arlington, Arlington Heights, Illinois
  - John H. Stroger, Jr., Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Elmhurst Memorial Hospital, Lombard, Illinois
  - Oncology Specialists, S.C., Niles, Illinois
  - US Oncology - Cancer Care & Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Orchard Research, Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - US Oncology - Cancer Care & Hematology Specialists of Chicagoland - Winfield, Winfield, Illinois
  - St. Francis Cancer Research, Beech Grove, Indiana
  - Center for Cancer Care @ Goshen Health Systems, Goshen, Indiana
  - Indiana University Cancer Center Clinical Research Office, Indianapolis, Indiana
  - Cancer Care Partners, LLC, Mishawaka, Indiana
  - Cancer Care Center, Inc., New Albany, Indiana
  - McFarland Clinic, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Iowa Blood and Cancer Care of PCI, Cedar Rapids, Iowa
  - Covenant Clinic, Waterloo, Iowa
  - Cancer Center of Kansas, PA, Wichita, Kansas
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Western Maryland Health System, Inc., Cumberland, Maryland
  - Alliance Hematology Oncology, PA, Westminster, Maryland
  - Capecod Hospital / Davenport Mugar Cancer Center, Hyannis, Massachusetts
  - Fallon Clinic, Worcester, Massachusetts
  - Michigan State University / McLaren Regional Medical Center, Flint, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Park Nicollet Institute Metro - MN CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Institute - Louisiana Ave., Saint Louis Park, Minnesota
  - US Oncology - University of Tennessee Cancer Institute - Southaven, Southaven, Mississippi
  - US Oncology - Missouri Cancer Associates, Columbia, Missouri
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - St. John's Medical Research Institute, Springfield, Missouri
  - Hematology Oncology Consultants, Inc., St Louis, Missouri
  - Montana Cancer Institute Foundation, Missoula, Montana
  - Nebraska Hematology Oncology, PC, Lincoln, Nebraska
  - Southeast Nebraska Hematology & Oncology Consultants, PC, Lincoln, Nebraska
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - VA Sierra Nevada Healthcare System, Reno, Nevada
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Drs. Forte, Schleider, Attas & Condemi, PA, Englewood, New Jersey
  - Charles Farber, MD, Morristown, New Jersey
  - Hematology Oncology of Northern New Jersey, Morristown, New Jersey
  - Steeplechase Cancer Center, Somerville, New Jersey
  - Samuel S Stratton VAMC, Albany, New York
  - Hematology Oncology Associates of Western Suffolk, Bay Shore, New York
  - Eduardo Saponara, MD, Bronxville, New York
  - Jonah Cancer Care Center & ECMC, Buffalo, New York
  - Broome Oncology, Johnson City, New York
  - SUNY Upstate Medical University - Adult Program, Syracuse, New York
  - Bronx River Medical Associates, The Bronx, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - US Oncology - Cancer Centers of North Carolina - Cary, Cary, North Carolina
  - US Oncology - Cancer Centers of North Carolina - Macon, Raleigh, North Carolina
  - US Oncology - Cancer Centers of North Carolina - Falls, Raleigh, North Carolina
  - Legacy Pharma Research, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Cancer Research Office, Akron, Ohio
  - Gabrail Cancer Center Research, Canton, Ohio
  - Mid Ohio Oncology / Hematology, Inc., Columbus, Ohio
  - Hematology Oncology Center, Inc., Elyria, Ohio
  - US Oncology - Willamette Valley Cancer Institute - Eugene, Eugene, Oregon
  - US Oncology - Northwest Cancer Specialists, PC - Portland - Hoyt, Portland, Oregon
  - US Oncology - Northwest Cancer Specialists, PC - Portland - Barnes, Portland, Oregon
  - US Oncology - Northwest Cancer Specialists, PC - Portland - Broadway, Portland, Oregon
  - US Oncology - Willamette Valley Cancer Institute - Springfield, Springfield, Oregon
  - US Oncology - Northwest Cancer Specialists, PC - Tualatin, Tualatin, Oregon
  - Oncology Hematology of Lehigh Valley, Bethlehem, Pennsylvania
  - Consultants in Medical Oncology and Hematology, PC, Drexel Hill, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Andrews and Patel Associates, Harrisburg, Pennsylvania
  - US Oncology - Medical Oncology Associates (Nahar), Kingston, Pennsylvania
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - Berks Hematology Oncology Associates, Reading, Pennsylvania
  - Hematology & Oncology Associates of Rhode Island, Cranston, Rhode Island
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - South Carolina Oncololgy Associates, PA, Columbia, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - Butternut, Greenville, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - West Faris, Greenville, South Carolina
  - US Oncology - Cancer Centers of the Carlinas - Eastside, Greenville, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Sanford Clinic, Sioux Falls, South Dakota
  - US Oncology - University of Tennessee Cancer Institute - Bartlett, Bartlett, Tennessee
  - Family Cancer Center, PLLC, Collierville, Tennessee
  - US Oncology - University of Tennessee Cancer Institute - Germantown, Germantown, Tennessee
  - US Oncology - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - SCRI, Nashville, Tennessee
  - US Oncology - Texas Cancer Center - Abilene (South), Abilene, Texas
  - US Oncology - Texas Oncology, PA - Amarillo, Amarillo, Texas
  - US Oncology - Texas Oncology - Arlington South, Arlington, Texas
  - US Oncology - Texas Oncology, PA - Bedford, Bedford, Texas
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Scott & White Clinic, College Station, Texas
  - South Texas Institute of Cancer, Corpus Christi, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - US Oncology - Texas Oncology, PA - Dallas, Dallas, Texas
  - US Oncology - El Paso Cancer Treatment Center - West, El Paso, Texas
  - US Oncology - El Paso Cancer Treatment Center, El Paso, Texas
  - US Oncology - Texas Oncology, PA - Fort Worth, Fort Worth, Texas
  - US Oncology - Southwest Fort Worth Cancer Center, Fort Worth, Texas
  - US Oncology - Texas Oncology - Grapevine, Grapevine, Texas
  - Oncology Consultants, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - US Oncology - San Antonio Tumor & Blood Clinic - Kerrville, Kerrville, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - US Oncology - Longview Cancer Center, Longview, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - US Oncology - Texas Oncology - McAllen, McAllen, Texas
  - US Oncology - Texas Oncology - Mesquite, Mesquite, Texas
  - US Oncology - Allison Cancer Center, Midland, Texas
  - US Oncology - Texas Oncology - Paris, Paris, Texas
  - US Oncology - Cancer Care Centers of South Texas, San Antonio, Texas
  - US Oncology - San Antonio Tumor & Blood Clinic - M. Oak, San Antonio, Texas
  - US Oncology - Texas Oncology - Sherman, Sherman, Texas
  - Scott & White Healthcare Department of Research, Temple, Texas
  - ETMC dba Blood and Cancer Center - East Texas, Tyler, Texas
  - ETMC dba Tyler Hematology Oncology, Tyler, Texas
  - US Oncology - Texas Oncology - Tyler, Tyler, Texas
  - US Oncology - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - US Oncology - Texas Oncology - Weslaco, Weslaco, Texas
  - US Oncology - Texoma Cancer Center, Wichita Falls, Texas
  - Central Utah Clinic, American Fork, Utah
  - Northern Utah Associates, Ogden, Utah
  - US Oncology - Arlington Fairfax Hematology Oncology, Arlington, Virginia
  - US Oncology - Onc and Hem Assoc of Southwest VA, Inc - Christiansburg, Christiansburg, Virginia
  - US Oncology - Fairfax Northern VA Hem-Onc PC, Fairfax, Virginia
  - US Oncology - Fairfax - Northern Virginia Hematology-Oncology, PC - Gainesville, Gainesville, Virginia
  - US Oncology - Fairfax - Northern Virginia Hem-Onc, PC - Leesburg, Leesburg, Virginia
  - US Oncology - Onc and Hem Assoc of Southwest VA, Inc - Low Moor, Low Moor, Virginia
  - US Oncology - Onc and Hem Assoc of Southwest VA, Inc - Roanoke, Roanoke, Virginia
  - US Oncology - Onc and Hem Assoc of Southwest VA, Inc - Salem, Salem, Virginia
  - US Oncology - Shenandoah Oncology - Winchester, Winchester, Virginia
  - US Oncology - Fairfax - Northern Virginia Hem-Onc, PC - Woodbridge, Woodbridge, Virginia
  - US Oncology - Onc and Hem Assoc of Southwest VA, Inc - Wytheville, Wytheville, Virginia
  - Peace Health Medical Group, Bellingham, Washington
  - US Oncology - Puget Sound Cancer Center - Edmonds, Edmonds, Washington
  - Providence Everett Medical Center, Everett, Washington
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - US Oncology - Puget Sound Cancer Center - Seattle, Seattle, Washington
  - US Oncology - Cancer Care Northwest - Sherman, Spokane, Washington
  - Medical Oncology Associates PS, Spokane, Washington
  - US Oncology - Cancer Care Northwest - Holland, Spokane, Washington
  - US Oncology - Cancer Care Northwest - Mission, Spokane, Washington
  - US Oncology - Northwest Cancer Specialists, PC - Vancouver - 136th St., Vancouver, Washington
  - US Oncology - Northwest Cancer Specialists, PC - Vancouver - 134th St, Vancouver, Washington
  - Providence St. Mary Regional Cancer Center, Walla Walla, Washington
  - US Oncology - Yakima Valley Memorial Hospital/North Star Lodge (Boyd), Yakima, Washington
  - St. Vincent Hospital/Green Bay Oncology, Green Bay, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin

REFERENCES:
- [Result] Pashos CL, Flowers CR, Kay NE, Weiss M, Lamanna N, Farber C, Lerner S, Sharman J, Grinblatt D, Flinn IW, Kozloff M, Swern AS, Street TK, Sullivan KA, Harding G, Khan ZM. Association of health-related quality of life with gender in patients with B-cell chronic lymphocytic leukemia. Support Care Cancer. 2013 Oct;21(10):2853-60. doi: 10.1007/s00520-013-1854-z. Epub 2013 Jun 8. PMID 23748484
- [Result] Mato A, Nabhan C, Kay NE, Weiss MA, Lamanna N, Kipps TJ, Grinblatt DL, Flinn IW, Kozloff MF, Flowers CR, Farber CM, Kiselev P, Swern AS, Sullivan K, Flick ED, Sharman JP. Real-world clinical experience in the Connect(R) chronic lymphocytic leukaemia registry: a prospective cohort study of 1494 patients across 199 US centres. Br J Haematol. 2016 Dec;175(5):892-903. doi: 10.1111/bjh.14332. Epub 2016 Nov 8. PMID 27861736
- [Result] Nabhan C, Mato A, Flowers CR, Grinblatt DL, Lamanna N, Weiss MA, Davids MS, Swern AS, Bhushan S, Sullivan K, Flick ED, Kiselev P, Sharman JP. Characterizing and prognosticating chronic lymphocytic leukemia in the elderly: prospective evaluation on 455 patients treated in the United States. BMC Cancer. 2017 Mar 16;17(1):198. doi: 10.1186/s12885-017-3176-x. PMID 28302090
- [Result] Mato A, Nabhan C, Kay NE, Lamanna N, Kipps TJ, Grinblatt DL, Flowers CR, Farber CM, Davids MS, Kiselev P, Swern AS, Bhushan S, Sullivan K, Flick ED, Sharman JP. Prognostic Testing Patterns and Outcomes of Chronic Lymphocytic Leukemia Patients Stratified by Fluorescence In Situ Hybridization/Cytogenetics: A Real-world Clinical Experience in the Connect CLL Registry. Clin Lymphoma Myeloma Leuk. 2018 Feb;18(2):114-124.e2. doi: 10.1016/j.clml.2017.11.010. Epub 2017 Dec 6. PMID 29352719
- [Result] Ahn IE, Farber CM, Davids MS, Grinblatt DL, Kay NE, Lamanna N, Mato A, Nabhan C, Kiselev P, Swern AS, Flick ED, Sullivan K, Sharman JP, Flowers CR. Early progression of disease as a predictor of survival in chronic lymphocytic leukemia. Blood Adv. 2017 Nov 28;1(25):2433-2443. doi: 10.1182/bloodadvances.2017011262. eCollection 2017 Nov 28. PMID 29296893
- [Result] Flowers CR, Nabhan C, Kay NE, Mato A, Lamanna N, Farber CM, Davids MS, Kiselev P, Swern AS, Sullivan K, Flick ED, Sharman JP. Reasons for initiation of treatment and predictors of response for patients with Rai stage 0/1 chronic lymphocytic leukemia (CLL) receiving first-line therapy: an analysis of the Connect(R) CLL cohort study. Leuk Lymphoma. 2018 Oct;59(10):2327-2335. doi: 10.1080/10428194.2018.1427860. Epub 2018 Feb 7. PMID 29415595
- [Derived] Mato A, Nabhan C, Lamanna N, Kay NE, Grinblatt DL, Flowers CR, Farber CM, Davids MS, Swern AS, Sullivan K, Flick ED, Gressett Ussery SM, Gharibo M, Kiselev P, Sharman JP. The Connect CLL Registry: final analysis of 1494 patients with chronic lymphocytic leukemia across 199 US sites. Blood Adv. 2020 Apr 14;4(7):1407-1418. doi: 10.1182/bloodadvances.2019001145. PMID 32271900